CLINICAL TRIAL: NCT03878914
Title: A Multinational Prospective Study on the Duration of Steroid Therapy in Steroid Sensitive Nephrotic Syndrome
Brief Title: Steroid Sensitive Nephrotic Syndrome in Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated at all but one site because of the pandemic
Sponsor: Wayne State University (Other)
Collaborators: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Tej Mattoo, MD, Professor of Pediatrics, Wayne State University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1901002013
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Nephrotic Syndrome in Children
Keywords: Nephrotic sydrome; Steroid sensitive nephrotic syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two groups based on time to remission with initial standard dose of corticosteroids. Patients who respond within 10 days (Group A) will receive a total of 8 weeks of corticosteroid therapy whereas those who respond between 10 days to 28 days (Group B) will receive ≥12 weeks ((maximum of 16 weeks) of corticosteroid therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quick responders (Group A) (Experimental): Patients will be divided into two groups based on time to remission with initial standard dose of corticosteroids. Patients who respond within 10 days (Group A) will receive a total of 8 weeks of corticosteroid therapy whereas those who respond between 10 days to 28 days (Group B) will receive ≥12 weeks ((maximum of 16 weeks) of corticosteroid therapy.
  CORTICOSTEROID THERAPY FOR INITIAL EPISODE Group A (Total duration of therapy 8 weeks)
  * 60mg/m2/day or 2mg/kg/day (maximum 60mg) day for 2 weeks
  * 40mg/m2 or 1.5mg (maximum 40mg) every other day for 2 weeks.
  * Wean off in 4 weeks
  CORTICOSTEROID THERAPY FOR A RELAPSE
  * 60mg/m2/day or 2mg/kg/day (maximum 60mg) until remission
  * 40mg/m2 or 1.5mg (maximum 40mg) every other day for one week followed by continued weaning until discontinued in 6-8 weeks.
  Interventions: Drug: Corticosteroids
- Slow responders (Group B) (Active Comparator): CORTICOSTEROID THERAPY FOR INITIAL EPISODE Group B: (Total duration of therapy ≥ 12 weeks)
  * 60mg/m2/day or 2mg/kg/day (maximum 60mg) day for 4 weeks
  * 40mg/m2 or 1.5mg (maximum 40mg) every other day for 4 weeks.
  * Wean off in 4-6 weeks
  CORTICOSTEROID THERAPY FOR A RELAPSE
  * 60mg/m2/day or 2mg/kg/day (maximum 60mg) until remission
  * 40mg/m2 or 1.5mg (maximum 40mg) every other day for one week followed by continued weaning until discontinued in 6-8 weeks.
  Interventions: Drug: Corticosteroids

INTERVENTIONS:
Drug: Corticosteroids — Patients will be divided into two groups based on time to remission with initial standard dose of corticosteroids. Patients who respond within 10 days (Group A) will receive a total of 8 weeks of corticosteroid therapy whereas those who respond between 10 days to 28 days (Group B) will receive ≥12 weeks ((maximum of 16 weeks) of corticosteroid therapy.

SUMMARY:
Idiopathic nephrotic syndrome (INS) is one of the most common glomerular pathologies in children and corticosteroid therapy is its most effective treatment. The total duration of treatment ranges anywhere from two to six months, generally about 3 months. The main objective of our study is to test the feasibility of a shorter total duration (two months) of corticosteroid therapy in patients who show a quicker treatment response to the initial treatment.

DETAILED DESCRIPTION:
Idiopathic nephrotic syndrome (INS) is one of the most common glomerular pathologies in children and corticosteroid therapy is its most effective treatment. The main objective of our prospective, open-label, observational clinical cohort study is to test the feasibility of a shorter duration of corticosteroid therapy in patients who show a quicker treatment response. We hypothesize that the clinical outcomes in children with time to remission of ≤10 days and treated with only 8 weeks of corticosteroid therapy will not be significantly different as compared to those with time to remission of >10 days and treated with ≥12 weeks of standard corticosteroid therapy. Our specific aims are as follows: First, we will evaluate the time to first relapse after 8-week corticosteroid therapy in quick responders in comparison to the standard treatment of ≥12 weeks in slow responders. Second, we will assess the frequency of relapses during one year follow-up after completion of 8-week corticosteroid therapy in quick responders in comparison to the standard treatment of ≥12 weeks in slow responders. To complete the study successfully during the funding period of two years and to increase the generalizability of its results, the study will recruit 66 patients at six study participating sites in five countries, including U.S., India, China, Egypt, and Qatar. The sites have been carefully selected on the basis of their reputation, patient volume, research experience, and PI's personal rapport with the site investigators. The proposed study is innovative because it seeks a paradigm shift from 'one-size-fits-all' to an entirely new concept of individualized treatment duration based on "time to remission" with initial corticosteroid therapy. The proposed study is the first precision medicine initiative in the management of INS. The project is significant because of the potential to improve public health by decreasing the side effects of prolonged corticosteroid administration in about half of the patients diagnosed with INS. Our long-term objective is to develop additional novel therapeutic strategies to optimize the use of corticosteroids in the management of initial episode and relapses in children with INS.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 to <19 years
* Newly diagnosed INS
* Patient in remission with steroids
* Written informed consent/Assent for the study OR as required by the local IRB

Exclusion Criteria:

* Age < 1 year or ≥ 19 years
* Uncertainty about patient/parent adherence.
* Abnormal serum creatinine for patient age
* Steroid resistant nephrotic syndrome
* Any co-morbid condition that might require modification in treatment with steroids.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Time to first relapse. | 60-64 weeks
  The study will evaluate the time in weeks for patients to relapse after completion of initial treatment and if there is any difference between Group A and Group B.

SECONDARY OUTCOMES:
Number of relapses | 52 weeks
  Number of relapses per patient after completion of treatment.
Number of frequent relapses | 52 weeks
  Number of frequent relapses per patient after completion of treatment.
Number of patients with steroid dependence | 52 weeks
  Number of patients who show steroid dependence after completion of treatment.
Number of patients with late steroid resistance | 52 weeks
  Number of patients who show late steroid resistance after completion of treatment.
Cumulative steroid dose in two groups | 60 to 64 weeks
  The total dose of corticosteroids received in Group A patients versus Group B patients
Number of episodes of upper respiratory infection (URI) and other infections. | 52-weeks
  The total number of URI or other infections in Group A patients versus Group B patients after completion of treatment.
Weight profile | 60-64 weeks
  Weight profile in Group A patients versus Group B patients
Height Profile | 60-64 weeks
  Height profile in Group A patients versus Group B patients

CONTACTS AND LOCATIONS:
Overall Officials: Tej Mattoo, MD, Principal Investigator — Wayne State University
Locations (2):
- Wayne Pediatrics, Detroit, Michigan, United States
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Depending on available resources, we may share data without any patient identifier with the study site investigators as well as others who might be interested.

REFERENCES:
- [Background] Hahn D, Hodson EM, Willis NS, Craig JC. Corticosteroid therapy for nephrotic syndrome in children. Cochrane Database Syst Rev. 2015 Mar 18;2015(3):CD001533. doi: 10.1002/14651858.CD001533.pub5. PMID 25785660
- [Background] Hodson EM, Willis NS, Craig JC. Corticosteroid therapy for nephrotic syndrome in children. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD001533. doi: 10.1002/14651858.CD001533.pub4. PMID 17943754
- [Background] Yoshikawa N, Nakanishi K, Sako M, Oba MS, Mori R, Ota E, Ishikura K, Hataya H, Honda M, Ito S, Shima Y, Kaito H, Nozu K, Nakamura H, Igarashi T, Ohashi Y, Iijima K; Japanese Study Group of Kidney Disease in Children. A multicenter randomized trial indicates initial prednisolone treatment for childhood nephrotic syndrome for two months is not inferior to six-month treatment. Kidney Int. 2015 Jan;87(1):225-32. doi: 10.1038/ki.2014.260. Epub 2014 Jul 23. PMID 25054775
- [Background] Sinha A, Saha A, Kumar M, Sharma S, Afzal K, Mehta A, Kalaivani M, Hari P, Bagga A. Extending initial prednisolone treatment in a randomized control trial from 3 to 6 months did not significantly influence the course of illness in children with steroid-sensitive nephrotic syndrome. Kidney Int. 2015 Jan;87(1):217-24. doi: 10.1038/ki.2014.240. Epub 2014 Jul 16. PMID 25029428
- [Background] Lombel RM, Hodson EM, Gipson DS; Kidney Disease: Improving Global Outcomes. Treatment of steroid-resistant nephrotic syndrome in children: new guidelines from KDIGO. Pediatr Nephrol. 2013 Mar;28(3):409-14. doi: 10.1007/s00467-012-2304-8. Epub 2012 Oct 5. PMID 23052648
- [Background] Vivarelli M, Moscaritolo E, Tsalkidis A, Massella L, Emma F. Time for initial response to steroids is a major prognostic factor in idiopathic nephrotic syndrome. J Pediatr. 2010 Jun;156(6):965-971. doi: 10.1016/j.jpeds.2009.12.020. Epub 2010 Mar 10. PMID 20223477
- [Background] Constantinescu AR, Shah HB, Foote EF, Weiss LS. Predicting first-year relapses in children with nephrotic syndrome. Pediatrics. 2000 Mar;105(3 Pt 1):492-5. doi: 10.1542/peds.105.3.492. PMID 10699098
- [Background] Letavernier B, Letavernier E, Leroy S, Baudet-Bonneville V, Bensman A, Ulinski T. Prediction of high-degree steroid dependency in pediatric idiopathic nephrotic syndrome. Pediatr Nephrol. 2008 Dec;23(12):2221-6. doi: 10.1007/s00467-008-0914-y. Epub 2008 Jul 11. PMID 18618150
- [Background] Srivastava RN, Mayekar G, Anand R, Choudhry VP, Ghai OP, Tandon HD. Nephrotic syndrome in indian children. Arch Dis Child. 1975 Aug;50(8):626-30. doi: 10.1136/adc.50.8.626. PMID 973
- [Background] Elzouki AY, Amin F, Jaiswal OP. Primary nephrotic syndrome in Arab children. Arch Dis Child. 1984 Mar;59(3):253-5. doi: 10.1136/adc.59.3.253. PMID 6712274
- [Background] Sharples PM, Poulton J, White RH. Steroid responsive nephrotic syndrome is more common in Asians. Arch Dis Child. 1985 Nov;60(11):1014-7. doi: 10.1136/adc.60.11.1014. PMID 4073933
- [Background] Banh THM, Hussain-Shamsy N, Patel V, Vasilevska-Ristovska J, Borges K, Sibbald C, Lipszyc D, Brooke J, Geary D, Langlois V, Reddon M, Pearl R, Levin L, Piekut M, Licht CPB, Radhakrishnan S, Aitken-Menezes K, Harvey E, Hebert D, Piscione TD, Parekh RS. Ethnic Differences in Incidence and Outcomes of Childhood Nephrotic Syndrome. Clin J Am Soc Nephrol. 2016 Oct 7;11(10):1760-1768. doi: 10.2215/CJN.00380116. Epub 2016 Jul 21. PMID 27445165
- [Background] Mattoo TK, Mahmood MA, al-Harbi MS. Nephrotic syndrome in Saudi children clinicopathological study of 150 cases. Pediatr Nephrol. 1990 Sep;4(5):517-9. doi: 10.1007/BF00869837. PMID 2242321
- [Background] Bagga A, Hari P, Srivastava RN. Prolonged versus standard prednisolone therapy for initial episode of nephrotic syndrome. Pediatr Nephrol. 1999 Nov;13(9):824-7. doi: 10.1007/s004670050708. PMID 10603129
- [Background] Hiraoka M, Tsukahara H, Matsubara K, Tsurusawa M, Takeda N, Haruki S, Hayashi S, Ohta K, Momoi T, Ohshima Y, Suganuma N, Mayumi M; West Japan Cooperative Study Group of Kidney Disease in Children. A randomized study of two long-course prednisolone regimens for nephrotic syndrome in children. Am J Kidney Dis. 2003 Jun;41(6):1155-62. doi: 10.1016/s0272-6386(03)00346-9. PMID 12776266
- [Derived] Tang X, Shen Q, Rao J, Chen J, Fang X, Zhang Z, Grewal M, Mattoo T, Xu H. Duration of initial prednisolone therapy for first episode of childhood nephrotic syndrome based on time to response. Front Pediatr. 2022 Nov 2;10:1043285. doi: 10.3389/fped.2022.1043285. eCollection 2022. PMID 36405821